CLINICAL TRIAL: NCT01977118
Title: Phase 2/3 Study of Use of Streptokinase for Enhancement of Percutaneous Drainage of Pancreatic Necrosis
Brief Title: Use of Streptokinase for Enhancement of Percutaneous Drainage of Pancreatic Necrosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajesh Gupta, Additional Professor, Division of Surgical Gastroenterology, Department of General Surgery, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NK/1180/M.CH
Record Dates: First submitted 2013-10-23; First posted 2013-11-06 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Acute Pancreatitis
Keywords: Streptokinase; Percutaneous catheter drainage; Pancreatic necrosis; peripancreatic necrosis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing | interventions — Streptokinase

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B [streptokinase] (Experimental): 50000U of injection streptokinase dissolved in 100ml of normal saline instilled in to the pancreatic and/or peripancreatic collections via the percutaneous catheters and clamped for 2 hours. After release of clamp, cavity will be irrigated with 100-500ml of normal saline. This procedure will be done thrice daily for five days
  Interventions: Drug: streptokinase
- Group A [placebo] (Placebo Comparator): 100 ml of normal saline will be instilled through percutaneous catheters in the pancreatic and/or peripancreatic collections and clamped for 2 hours. After release of clamp, cavity will be irrigated with 100-500ml of saline. This procedure will be performed thrice daily for five days
  Interventions: Other: Saline irrigation

INTERVENTIONS:
Drug: streptokinase — 50000U of injection streptokinase dissolved in 100ml of diluent instilled in to the pancreatic and/or peripancreatic collections via percutaneous catheters and clamped for 2 hours in Streptokinase group. After release of clamp, cavity will be irrigated with 100-500ml of saline. This procedure will be performed thrice daily for five days.
  Arms: Group B [streptokinase]
Other: Saline irrigation — 100 ml of normal saline will be instilled through percutaneous catheters in the pancreatic and/or peripancreatic collections and clamped for 2 hours. After release of clamp, cavity will be irrigated with 100-500ml of saline. This procedure will be performed thrice daily for five days
  Arms: Group A [placebo]

SUMMARY:
Around 20 per cent of patients with acute pancreatitis develop pancreatic or peripancreatic necrosis with or without peripancreatic collection.

Percutaneous catheter drainage successfully drains the liquefied component of pancreatic necrosis while the solid component still remains undrained. This infected solid component of pancreatic necrosis is probably responsible for failure of percutaneous catheter drainage which demands surgical debridement.

Streptokinase is a protein secreted by several species of streptococci which can bind and activate human plasminogen.

In the present study investigators plan to instill streptokinase locally in to the collections of patients with severe acute pancreatitis via pigtail catheter inorder to liquefy the solid necrotic component and analyze whether it hastens the drainage and thereby delays or obviates the need for necrosectomy.

DETAILED DESCRIPTION:
Around 20 per cent of patients with acute pancreatitis develop pancreatic or peripancreatic necrosis with or without peripancreatic collections. Sterile necrosis can generally be managed conservatively and the mortality rate is relatively low (12 per cent). Approximately 30 (range 14-62) per cent of patients with necrotizing pancreatitis, however, develop secondary infections of peripancreatic fluid collection which is associated with sepsis and organ failure and is an indication for intervention1.

Until recently, the first-choice intervention in patients with infected necrotizing pancreatitis or sterile necrosis with clinical deterioration (multiple organ failure) has been open surgical necrosectomy. This approach is associated with considerable morbidity (34-95 per cent) and mortality (11-39 per cent). In 1998, Freeny and colleagues10 first described a consecutive series of patients with infected pancreatic necrosis who were treated primarily with imaging-guided percutaneous catheter drainage (PCD), as an alternative to primary surgical necrosectomy. The rationale for PCD was to drain the infected fluid under tension and gain time to improve organ function of these critically ill patients and thereby delay or avoid surgical necrosectomy. In their retrospective cohort study, PCD was successful in postponing surgical intervention for a median of 4 weeks and even obviated the need for surgical necrosectomy in almost half of the patients. In addition, PCD seems technically feasible in the vast majority of patients with necrotizing pancreatitis.

In clinical experience, investigators have found that PCD successfully drains the liquefied component of pancreatic necrosis while the solid component still remains undrained. This infected solid component of pancreatic necrosis is probably responsible for failure of PCD which demands surgical debridement.

Streptokinase is a protein secreted by several species of streptococci which can bind and activate human plasminogen. It is primarily used in clinical practice intravenously as an effective thrombolytic agent in cases of myocardial infarction and pulmonary thromboembolism.

The earliest reports on intracavitatory use of Streptokinase and other fibrinolytics were for empyemas. Later because of beneficial results, their intracavitatory use was extended to other conditions like liver, retroperitoneal and peritoneal abscesses.

In a phase II study, intracavitatory urokinase has shown to facilitate percutaneous drainage significantly reduce hospital stay and costs of percutaneous drainage of intra abdominal, retroperitoneal abscesses.

In the present study investigators plan to instill streptokinase locally in to the collections of patients with severe acute pancreatitis via pigtail catheter inorder to liquefy the solid necrotic component and analyze whether it hastens the drainage and thereby delays or obviates the need for necrosectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe acute pancreatitis managed by percutaneous catheter drainage

Exclusion Criteria:

* An acute intra abdominal event (perforation of hollow viscus, bleeding, or abdominal compartment syndrome) before or after PCD insertion.
* Previous drainage or surgical necrosectomy for infected pancreatic necrosis (ERCP with or without papillotomy is allowed.)
* Previous exploratory laparotomy for acute abdomen and diagnosis of pancreatitis during laparotomy
* Patients who are allergic to streptokinase.
* Patients with deranged coagulation profile.
* Patients with recent history of cerebrovascular accident [< 2 months], intracranial or intraspinal surgery, uncontrolled hypertension, intracranial neoplasm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sepsis reversal | From date of randomization until the date of necrosectomy, discharge or death from any cause, whichever came first, assessed upto 1 month
Mortality | From the date of randomization until last follow up after discharge, assessed up to 1 month

SECONDARY OUTCOMES:
Length of intensive care unit (ICU) and hospital stay | From date of randomization until the date of discharge or death from any cause, whichever came first, assessed upto 1 month
Proportion of patients requiring surgical necrosectomy | From date of randomization until the date of discharge or death from any cause, whichever came first, assessed upto 1 month
Number and size of catheters required | From date of first pigtail insertion until the date of necrosectomy, discharge or death from any cause, whichever came first, assessed upto 1 month
Number of interventions required | From date of first pigtail insertion until the date of necrosectomy, discharge or death from any cause, whichever came first, assessed upto 1 month
Catheter-related complications | From date of first pigtail insertion until the date of necrosectomy, discharge or death from any cause, whichever came first, assessed upto 1 month
Streptokinase related complications | From date of randomization until the date of necrosectomy, discharge or death from any cause, whichever came first, assessed upto 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Gupta, M.Ch., Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India